CLINICAL TRIAL: NCT00866697
Title: A Phase III Study to Evaluate the Efficacy and Safety of Pazopanib Monotherapy Versus Placebo in Women Who Have Not Progressed After First Line Chemotherapy for Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Efficacy and Safety of Pazopanib Monotherapy After First Line Chemotherapy in Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 110655; 2008-004672-50 (EudraCT Number); CPZP034C2301 (Other: Novartis)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer
Keywords: fallopian tube cancer; pazopanib; anti-angiogenesis; ovarian cancer; primary peritoneal cancer; tyrosine kinase inhibitors; gynecologic cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): matched placebo tablet administered orally once daily for up to 24 months
  Interventions: Drug: Placebo
- Pazopanib (Experimental): Pazopanib tablet administered orally at 800 mg once daily for up to 24 months
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 800 mg tablet daily for 104 weeks (24 months)
  Arms: Pazopanib
Drug: Placebo — Matching placebo 800 mg tablet daily, for 104 weeks (24 months).
  Arms: Placebo

SUMMARY:
This was a study to determine whether therapy with pazopanib was effective and safe in women with epithelial ovarian, fallopian tube, or primary peritoneal cancer whose cancer had not progressed on first line chemotherapy.

DETAILED DESCRIPTION:
This was a randomized, two-arm, placebo controlled, double-blind, multicenter, intergroup Phase III study in women with non-bulky FIGO (International Federation of Gynecology and Obstetrics) Stage II - IV ovarian, fallopian tube, or primary peritoneal cancer that had not progressed (i.e., complete response (CR), partial response (PR), stable disease (SD) after completing their first-line chemotherapy for advanced ovarian cancer. Approximately 900 subjects were to be enrolled into the study. Study was closed following 3rd overall survival (OS) interim analysis as planned per protocol, which confirmed futility.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* At least 18 years old.
* Histologically confirmed, FIGO stage II-IV epithelial ovarian, fallopian tube or primary peritoneal carcinoma that was treated with surgical debulking and at least five cycles of platinum-taxane doublet chemotherapy.
* Study randomization at least 3 weeks and not more than 12 weeks from the date of the last chemotherapy dose, and all major toxicities from the previous chemotherapy must have resolved.
* No evidence of disease progression
* ECOG status of 0 or 2
* Able to swallow and retain oral medication.
* Adequate hematologic, hepatic, and renal system function as follows:

Hematologic

* Absolute neutrophil count (ANC) at least 1.5 X 10^9/L
* Hemoglobin at least 9 g/dL (or 5.59 mmol/L)
* Platelets at least 100 X 10^9/L
* Prothrombin time (PT) or international normalized ratio (INR) up to 1.2 X ULN
* Activated partial thromboplastin time (aPTT) up to 1.2 X ULN Hepatic
* Total bilirubin up to 1.5 X ULN
* AST and ALT up to 2.5 X ULN Renal
* Serum creatinine up to 1.5 mg/dL

Or, if greater than 1.5 mg/dL:

Calculated creatinine clearance at least 50 mL/min Urine Protein

* Urine protein is 0, trace, or +1 determined by dipstick urinalysis, or < 1.0 gram determined by 24- hour urine protein analysis.
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) OR childbearing potential, and agrees to use adequate contraception.

Exclusion Criteria:

* Either (a) bulky disease, or (b) any residual disease which in the opinion of the investigator will need imminent second-line therapy
* Synchronous primary endometrial carcinoma, or a past history of primary endometrial carcinoma, are excluded unless certain conditions are met.
* Clinically significant gastrointestinal abnormalities
* Prolongation of corrected QT interval (QTc) > 480 msecs
* History of any one or more cardiovascular conditions within the past 6 months prior to randomization
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Symptomatic peripheral vascular disease

  * Class III or IV congestive heart failure
* Poorly controlled hypertension
* History of cerebrovascular accident (including transient ischemic attacks), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months prior to randomization
* Major surgery (including interval debulking) or trauma within 28 days, or minor surgical procedures within 7 days, prior to randomization, or has any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Hemoptysis within 6 weeks prior to randomization.
* Endobronchial metastases.
* Serious and/or unstable pre-existing medical (e.g., uncontrolled infection), psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Investigational or anti-VEGF anticancer therapy prior to study randomization.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib
* Invasive malignancies that showed activity of disease within 5 years prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2009-05-26 (Actual); Primary Completion 2012-07-08 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (246):
- United States (30):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Baldwin Park, California
  - Novartis Investigative Site, Bellflower, California
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Fontana, California
  - Novartis Investigative Site, Hayward, California
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Ontario, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Panorama City, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Roseville, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Santa Clara, California
  - Novartis Investigative Site, South San Francisco, California
  - Novartis Investigative Site, Vallejo, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Woodland Hills, California
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Morristown, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Annandale, Virginia
- Australia (13):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Wodonga, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Melbourne
- Austria (9):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Klagenfurt
  - Novartis Investigative Site, Korneuburg
  - Novartis Investigative Site, Krems
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Oberpullendorf
  - Novartis Investigative Site, Vienna
- Belgium (9):
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Duffel
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Libramont
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Ostend
- China (8):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Denmark (4):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Herning
  - Novartis Investigative Site, Koebenhavn Oe
- France (40):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bourg-en-Bresse
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Brive-la-Gaillarde
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Dax
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Mont-de-Marsan
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mougins
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perin Sur Mer
  - Novartis Investigative Site, Périgueux
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Suresnes
  - Novartis Investigative Site, Thonon-les-Bains
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (69):
  - Novartis Investigative Site, Esslingen am Neckar, Baden-Wurttemberg
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Karlsruhe, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Mutlangen, Baden-Wurttemberg
  - Novartis Investigative Site, Reutlingen, Baden-Wurttemberg
  - Novartis Investigative Site, Schwäbisch Hall, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Bayreuth, Bavaria
  - Novartis Investigative Site, Coburg, Bavaria
  - Novartis Investigative Site, Deggendorf, Bavaria
  - Novartis Investigative Site, Ebersberg, Bavaria
  - Novartis Investigative Site, Eggenfelden, Bavaria
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Schweinfurt, Bavaria
  - Novartis Investigative Site, Darmstadt, Hesse
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Fulda, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Lich, Hesse
  - Novartis Investigative Site, Limburg an der Lahn, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Offenbach, Hesse
  - Novartis Investigative Site, Wiesbaden, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Cuxhaven, Lower Saxony
  - Novartis Investigative Site, Georgsmarienhütte, Lower Saxony
  - Novartis Investigative Site, Gifhorn, Lower Saxony
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Hildesheim, Lower Saxony
  - Novartis Investigative Site, Leer, Lower Saxony
  - Novartis Investigative Site, Lüneburg, Lower Saxony
  - Novartis Investigative Site, Oldenburg, Lower Saxony
  - Novartis Investigative Site, Salzgitter, Lower Saxony
  - Novartis Investigative Site, Wolfsburg, Lower Saxony
  - Novartis Investigative Site, Greifswald, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Detmold, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Neuss, North Rhine-Westphalia
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Viersen, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Trier, Rhineland-Palatinate
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzg, Saxony
  - Novartis Investigative Site, Radebeul, Saxony
  - Novartis Investigative Site, Zwickau, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Quedlinburg, Saxony-Anhalt
  - Novartis Investigative Site, Salzwedel, Saxony-Anhalt
  - Novartis Investigative Site, Flensburg, Schleswig-Holstein
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Gera, Thuringia
  - Novartis Investigative Site, Nordhausen, Thuringia
  - Novartis Investigative Site, Suhl, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
- Ireland (3):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Waterford
  - Novartis Investigative Site, Wilton, Cork
- Italy (21):
  - Novartis Investigative Site, Bari, Apulia
  - Novartis Investigative Site, Potenza, Basilicate
  - Novartis Investigative Site, Avellino, Campania
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Bologna, Emilia-Romagna
  - Novartis Investigative Site, Carpi (MO), Emilia-Romagna
  - Novartis Investigative Site, Faenza (RA), Emilia-Romagna
  - Novartis Investigative Site, Reggio Emilia, Emilia-Romagna
  - Novartis Investigative Site, Aviano (PN), Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Brescia, Lombardy
  - Novartis Investigative Site, Como, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Monza, Lombardy
  - Novartis Investigative Site, Sondrio, Lombardy
  - Novartis Investigative Site, Varese, Lombardy
  - Novartis Investigative Site, Campobasso, Molise
  - Novartis Investigative Site, Turin, Piedmont
  - Novartis Investigative Site, Palermo, Sicily
  - Novartis Investigative Site, Perugia, Umbria
  - Novartis Investigative Site, Vicenza, Veneto
- Japan (11):
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Hokkaido
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Numakunai
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Tottori
- Norway (4):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Tromsø
- South Korea (3):
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Kangnam-Ku ,Seoul
  - Novartis Investigative Site, Seoul
- Spain (15):
  - Novartis Investigative Site, Alcorcon (Madrid)
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Cartagena (Murcia)
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Elche
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia (El Palmar)
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Sabadell (Barcelona)
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Terrassa
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Sweden (4):
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Vergote I, du Bois A, Floquet A, Rau J, Kim JW, Del Campo JM, Friedlander M, Pignata S, Fujiwara K, Colombo N, Mirza MR, Monk BJ, Tsibulak I, Calvert PM, Herzog TJ, Hanker LC, Meunier J, Lee JY, Bologna A, Carrasco-Alfonso MJ, Harter P. Overall survival results of AGO-OVAR16: A phase 3 study of maintenance pazopanib versus placebo in women who have not progressed after first-line chemotherapy for advanced ovarian cancer. Gynecol Oncol. 2019 Nov;155(2):186-191. doi: 10.1016/j.ygyno.2019.08.024. Epub 2019 Sep 10. PMID 31519320
- [Derived] Friedlander M, Rau J, Lee CK, Meier W, Lesoin A, Kim JW, Poveda A, Buck M, Scambia G, Shimada M, Hilpert F, King MT, Debruyne P, Bologna A, Malander S, Monk BJ, Petru E, Calvert P, Herzog TJ, Barrett C, du Bois A. Quality of life in patients with advanced epithelial ovarian cancer (EOC) randomized to maintenance pazopanib or placebo after first-line chemotherapy in the AGO-OVAR 16 trial. Measuring what matters-patient-centered end points in trials of maintenance therapy. Ann Oncol. 2018 Mar 1;29(3):737-743. doi: 10.1093/annonc/mdx796. PMID 29267856
- [Derived] Pulford DJ, Harter P, Floquet A, Barrett C, Suh DH, Friedlander M, Arranz JA, Hasegawa K, Tada H, Vuylsteke P, Mirza MR, Donadello N, Scambia G, Johnson T, Cox C, Chan JK, Imhof M, Herzog TJ, Calvert P, Wimberger P, Berton-Rigaud D, Lim MC, Elser G, Xu CF, du Bois A. Communicating BRCA research results to patients enrolled in international clinical trials: lessons learnt from the AGO-OVAR 16 study. BMC Med Ethics. 2016 Oct 21;17(1):63. doi: 10.1186/s12910-016-0144-y. PMID 27769273
- [Derived] Kim JW, Mahner S, Wu LY, Shoji T, Kim BG, Zhu JQ, Takano T, Park SY, Kong BH, Wu Q, Wang KL, Ngan HY, Liu JH, Wei LH, Mitrica I, Zhang P, Crescenzo R, Wang Q, Cox CJ, Harter P, du Bois A. Pazopanib Maintenance Therapy in East Asian Women With Advanced Epithelial Ovarian Cancer: Results From AGO-OVAR16 and an East Asian Study. Int J Gynecol Cancer. 2018 Jan;28(1):2-10. doi: 10.1097/IGC.0000000000000602. PMID 26588236
- [Derived] Floquet A, Vergote I, Colombo N, Fiane B, Monk BJ, Reinthaller A, Calvert P, Herzog TJ, Meier W, Kim JW, del Campo JM, Friedlander M, Pisano C, Isonishi S, Crescenzo RJ, Barrett C, Wang K, Mitrica I, du Bois A. Progression-free survival by local investigator versus independent central review: comparative analysis of the AGO-OVAR16 Trial. Gynecol Oncol. 2015 Jan;136(1):37-42. doi: 10.1016/j.ygyno.2014.11.074. Epub 2014 Nov 28. PMID 25434635
- [Derived] du Bois A, Floquet A, Kim JW, Rau J, del Campo JM, Friedlander M, Pignata S, Fujiwara K, Vergote I, Colombo N, Mirza MR, Monk BJ, Kimmig R, Ray-Coquard I, Zang R, Diaz-Padilla I, Baumann KH, Mouret-Reynier MA, Kim JH, Kurzeder C, Lesoin A, Vasey P, Marth C, Canzler U, Scambia G, Shimada M, Calvert P, Pujade-Lauraine E, Kim BG, Herzog TJ, Mitrica I, Schade-Brittinger C, Wang Q, Crescenzo R, Harter P. Incorporation of pazopanib in maintenance therapy of ovarian cancer. J Clin Oncol. 2014 Oct 20;32(30):3374-82. doi: 10.1200/JCO.2014.55.7348. Epub 2014 Sep 15. PMID 25225436

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching placebo once daily for a maximum of 24 months.
- Pazopanib 800 mg: Participants received pazopanib 800 milligrams (mg) once daily for a maximum of 24 months.
Period: Overall Study
Arm/Group | Placebo | Pazopanib 800 mg
Started | 468 | 472
Completed (Death) | 254 | 244
Not Completed | 214 | 228
Not completed — Study closed/terminated | 156 | 138
Not completed — Lost to Follow-up | 22 | 28
Not completed — Physician Decision | 3 | 5
Not completed — Withdrawal by Subject | 33 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pazopanib 800 mg | Total
Number analyzed (Participants) | 468 | 472 | 940
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (10.83) | 55.8 (10.54) | 56.3 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 468 | 472 | 940
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 2 | 3
  American Indian or Alaska Native | 1 | 1 | 2
  Central/South Asian Heritage (Her) | 1 | 0 | 1
  Japanese/East Asian Her/South East Asian Her | 102 | 106 | 208
  White | 363 | 363 | 726

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Progression-free Survival (PFS)
Description: PFS is the interval between the date of randomization and the date of progression, defined by Response Evaluation Criteria in Solid Tumors (RECIST), or death due to any cause. Per RECIST, for target lesions (TLs), disease progression (PD) is defined as >=20% increase in the sum of the longest diameters (LD) of TLs, taking as a reference, the smallest sum LD recorded since the treatment started or the appearance of >=1 new lesions. For non-target lesions (NTLs), PD is defined as the appearance of >=1 new lesions and/or unequivocal progression of existing NTLs. Participants (par.) who did not progress/die were censored at the date of last adequate assessment (LAA). Par. who started a new anti-cancer therapy (ACT) prior to radiological progression/death were censored at the date of LAA prior to the new ACT. Par. who progressed/died after an extended period (>=12 months) without adequate assessment (AA) were censored at the date of their last visit with AA prior to progression/death.
Time Frame: From the date of randomization until the date of progression or death due to any cause (median time of follow-up was 17.9 months for pazopanib and 12.3 months for placebo)
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 468 | 472
months | 12.3 [11.8 to 17.7] | 17.9 [15.9 to 21.8]
Statistical Analysis 1: Comparison: Placebo vs Pazopanib 800 mg; Test type: Superiority or Other; p = 0.0021, Log Rank — The P-value from the stratified log-rank test was adjusted for the two stratification factors; Hazard Ratio (HR) = 0.766, 95% CI 2-sided [0.643 to 0.911] — The Hazard Ratio was estimated using a Pike estimator

2. Secondary Outcome: Overall Survival - Median
Description: Overall surival is defined as the interval between the date of randomization and the date of death due to any cause. For participants who did not die, the time to death was censored at the time of last contact.
Time Frame: From the date of randomization until the date of death due to any cause up to approximately 25 months
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 468 | 472
months | 64.0 [56.0 to 75.7] | 59.1 [53.5 to 71.6]
Statistical Analysis 1: Comparison: Placebo vs Pazopanib 800 mg; Test type: Superiority; p = 0.6431, Log Rank; Stratified Log-Rank P-Value; Hazard Ratio (HR) = 0.960, 95% CI 2-sided [0.805 to 1.145] — The HR was estimated using a Pike estimator. CIs were estimated using the Brookmeyer-Crowley method

3. Secondary Outcome: Overall Survival: Number of Participants Experiencing Death
Description: as for outcome 2
Time Frame: From the date of randomization until the date of death due to any cause up to approximately 25 months
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 468 | 472
participants
  deaths | 253 | 241
  censored, follow up ended (no deaths) | 215 | 231

4. Secondary Outcome: Progression-free Survival Per Gynecologic Cancer Intergroup (GCIG) Criteria
Description: Progression-free survival by GCIG criteria is defined as the time from the date of randomization to the earliest date of disease progression per GCIG criteria or death due to any cause. Progression is defined according to RECIST but can also be based upon serum CA-125. Progression or recurrence based on serum CA-125 levels are defined on the basis of a progressive serial elevation of serum CA-125, according to the following criteria: (1) participants (par.) with elevated CA-125 pretreatment and normalization of CA-125 must show evidence of CA-125 >=2x the upper normal limit (UNL) on two occasions at least one week apart or; (2) par. with elevated CA-125 pretreatment, which never normalizes, must show evidence of CA-125 >=2x the nadir value on two occasions at least one week apart or; (3) par. with CA-125 in the normal range pretreatment must show evidence of CA-125 >=2x the UNL on two occasions at least one week apart.
Time Frame: From the date of randomization until the date of progression per GCIG criteria or death due to any cause (median time of follow-up was 16.8 months for pazopanib and 11.9 months for placebo)
Population: Intent-to-Treat (ITT) Population: all randomized participants.
  For participants who did not progress or die, progression-free survival was censored at the time of the last adequate disease assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 468 | 472
months | 11.9 [10.6 to 14.9] | 16.8 [12.6 to 18.1]

5. Secondary Outcome: 3-year Progression-free Survival
Description: 3-year progression-free survival is defined as the percentage of participants who are progression-free at 3 years from randomization. Progression-free survival is defined as the time from the date of randomization to the earliest date of disease progression (defined by RECIST) or death due to any cause. Per RECIST, for target lesions, disease progression (PD) is defined as at least a 20% increase in the sum of the longest diameters (LD) of target lesions, taking as a reference, the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions, PD is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 3 years after randomization
Population: Intent-to-Treat (ITT) Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 468 | 472
percentage of participants | NA — At the time of data cut-off, only one participant had more than 3 years of follow-up; therefore, 3-year progression-free survival could not be estimated. | NA — At the time of data cut-off, only one participant had more than 3 years of follow-up; therefore, 3-year progression-free survival could not be estimated.

6. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer (EORTC) QLQ-C30 Global Health Status Score on Day 1 of Week 13 and Months 7, 10, 13, 16, and 25
Description: The EORTC QLQ-C30 is a self-reported, 30-item cancer-specific instrument that assesses 15 domains: 5 functional scales (physical, role, emotional, cognitive, and social functioning), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a global health status, or quality of life. Global health status is assessed using a 7-item Likert scale, ranging from 1 to 7 ("poor" to "excellent"). Participants were asked to respond to the following questions using the 7-item Likert scale: "How would you rate your overall health during the past week"; "How would you rate your overall quality of life during the past week?" Data are transformed to a scale ranging from 0 to 100. Higher scores represent better functioning (better quality of life). Mean changes from Baseline were calculated via mixed model-repeated measures analysis of covariance (ANCOVA).
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 393 | 293
scores on a scale
  Week 13 | 0.58 (0.821) | -3.82 (0.950)
  Month 7: number analyzed (Participants) | 316 | 223
  Month 7 | 0.95 (0.962) | -4.65 (1.139)
  Month 10: number analyzed (Participants) | 240 | 184
  Month 10 | 1.98 (0.972) | -4.28 (1.115)
  Month 13: number analyzed (Participants) | 190 | 140
  Month 13 | 0.65 (1.200) | -1.80 (1.398)
  Month 16: number analyzed (Participants) | 137 | 87
  Month 16 | 1.39 (1.370) | 0.96 (1.702)
  Month 25: number analyzed (Participants) | 92 | 53
  Month 25 | 3.86 (1.488) | -1.68 (1.934)

7. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Attitude to Disease/Treatment Functional Score on Day 1 of Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV (ovarian)-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses attitude to disease/treatment functional symptoms, among others. Participants were asked to indicate the extent to which they experienced attention to disease/treatment functional problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: How much has your disease been a burden to you?; How much has your treatment been a burden to you?; Were you worried about your future health? Data are transformed to a scale ranging from 0 to 100. Higher scores represent better functioning (better quality of life). Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 378 | 291
scores on a scale
  Week 13 | 9.92 (1.110) | 4.24 (1.263)
  Month 7: number analyzed (Participants) | 299 | 223
  Month 7 | 12.10 (1.203) | 4.94 (1.385)
  Month 10: number analyzed (Participants) | 228 | 185
  Month 10 | 14.31 (1.310) | 8.54 (1.467)
  Month 13: number analyzed (Participants) | 182 | 138
  Month 13 | 15.45 (1.388) | 10.07 (1.589)
  Month 16: number analyzed (Participants) | 133 | 88
  Month 16 | 15.81 (1.668) | 13.25 (2.013)
  Month 25: number analyzed (Participants) | 90 | 54
  Month 25 | 16.50 (2.021) | 5.72 (2.565)

8. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Body Image Functional Score on Day 1 of Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses body image symptoms, among others. Participants were asked to indicate the extent to which they experienced body image problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: Have you felt physically less attractive as a result of your disease or treatment?; Have you been dissatisfied with your body? Data are transformed to a scale ranging from 0 to 100. Higher scores represent better functioning (better quality of life). Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 386 | 297
scores on a scale
  Week 13 | 7.18 (1.063) | 2.99 (1.210)
  Month 7: number analyzed (Participants) | 312 | 230
  Month 7 | 7.88 (1.141) | 4.26 (1.319)
  Month 10: number analyzed (Participants) | 236 | 190
  Month 10 | 8.12 (1.319) | 4.65 (1.482)
  Month 13: number analyzed (Participants) | 187 | 145
  Month 13 | 8.54 (1.421) | 4.34 (1.616)
  Month 16: number analyzed (Participants) | 133 | 91
  Month 16 | 7.68 (1.633) | 6.21 (1.941)
  Month 25: number analyzed (Participants) | 88 | 56
  Month 25 | 10.81 (1.856) | 3.10 (2.281)

9. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Peripheral Neuropathy (PN) Symptoms Score at Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses peripheral neuropathy symptoms, among others. Participants were asked to indicate the extent to which they experienced peripheral neuropathy symptoms or problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: Did you have tingling hands or feet?; Have you had numbness in your fingers or toes?; Have you felt weak in your arms or legs? Data are transformed to a scale from 0 to 100. Lower scores represent better health (fewer symptoms) for symptom scales. Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 388 | 297
scores on a scale
  Week 13 | -3.34 (1.038) | -5.22 (1.184)
  Month 7: number analyzed (Participants) | 301 | 226
  Month 7 | -6.12 (1.104) | -5.20 (1.270)
  Month 10: number analyzed (Participants) | 235 | 188
  Month 10 | -7.85 (1.209) | -5.11 (1.361)
  Month 13: number analyzed (Participants) | 188 | 140
  Month 13 | -8.76 (1.301) | -6.37 (1.499)
  Month 16: number analyzed (Participants) | 133 | 90
  Month 16 | -8.66 (1.456) | -8.65 (1.745)
  Month 25: number analyzed (Participants) | 91 | 55
  Month 25 | -9.47 (1.595) | -8.30 (2.010)

10. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Abdominal (AB)/Gastrointestinal (GI) Symptoms Score at Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses AB/GI symptoms, among others. Participants were asked to indicate the extent to which they experienced AB/GI symptoms or problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: Did you have abdominal pain?; Did you have a bloated feeling in your abdomen/stomach?; Did you have problems with your clothes feeling too tight?; Did you experience any change in bowel habit as a result of your disease or treatment?; Were you troubled by passing wind/gas/flatulence?; Have you felt full too quickly after beginning to eat?; Have you had indigestion/heartburn? Data are transformed to a scale from 0 to 100. Lower scores represent better health (fewer symptoms) for symptom scales. Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 388 | 289
scores on a scale
  Week 13 | 0.93 (0.673) | 6.62 (0.777)
  Month 7: number analyzed (Participants) | 308 | 225
  Month 7 | 2.36 (0.831) | 11.11 (0.967)
  Month 10: number analyzed (Participants) | 232 | 187
  Month 10 | 2.74 (0.957) | 11.33 (0.957)
  Month 13: number analyzed (Participants) | 187 | 141
  Month 13 | 3.64 (1.027) | 12.29 (1.181)
  Month 16: number analyzed (Participants) | 133 | 88
  Month 16 | 3.69 (1.251) | 8.11 (1.503)
  Month 25: number analyzed (Participants) | 91 | 54
  Month 25 | 3.82 (1.388) | 11.86 (1.762)

11. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Hormonal/Menopausal Symptoms Score at Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses hormonal/menopausal symptoms, among others. Participants were asked to indicate the extent to which they experienced hormonal/menopausal symptoms or problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: Did you have hot flashes?; Did you have night sweats? Data are transformed to a scale from 0 to 100. Lower scores represent better health (fewer symptoms) for symptom scales. Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 398 | 299
scores on a scale
  Week 13 | -0.86 (1.026) | -0.95 (1.177)
  Month 7: number analyzed (Participants) | 315 | 232
  Month 7 | -0.38 (1.185) | 1.29 (1.371)
  Month 10: number analyzed (Participants) | 239 | 189
  Month 10 | -2.17 (1.299) | 0.83 (1.470)
  Month 13: number analyzed (Participants) | 186 | 144
  Month 13 | -2.77 (1.396) | -0.74 (1.594)
  Month 16: number analyzed (Participants) | 136 | 91
  Month 16 | -0.41 (1.610) | 1.09 (1.920)
  Month 25: number analyzed (Participants) | 92 | 55
  Month 25 | -1.58 (1.798) | -0.68 (2.280)

12. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Sexuality Functional on Day 1 of Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses sexual functioning symptoms, among others. Participants were asked to indicate the extent to which they experienced sexual functioning problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: To what extent were you interested in sex?; To what extent were you sexually active?; If sexually active, to what extent was sex enjoyable for you?; If sexually active, did you have a dry vagina during sexual activity? Higher scores represent better functioning (better quality of life). Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA. Data were not analyzed due to low compliance (<50% at Baseline).
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: Data were not analyzed due to low compliance (<50% at Baseline).
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in QLQ-OV-28 Module Other Chemotherapy Side Effects (SE) Symptoms Score at Week 13 and Months 7, 10, 13, 16, and 25
Description: The OV-28 module is a 28-item addition to the EORTC QLQ-C30 that focuses on issues specific to ovarian cancer. It assesses other chemotherapy SE symptoms, among others. Participants were asked to indicate the extent to which they experienced other chemotherapy SE symptoms/problems in the week prior to assessment. Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) to the following questions: Have you lost any hair?; If yes, were you upset by the loss of your hair?; Did food/drink taste different from usual?; Did you have aches or pains in your muscles or joints?; Did you have problems with hearing?; Did you urinate frequently?; Have you had skin problems (e.g., itchy, dry)? Data are transformed to a scale from 0 to 100. Lower scores represent better health (fewer symptoms) for symptom scales. Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA. Data were not analyzed due to low compliance (<50% at Baseline).
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA. Data were not analyzed due to low compliance (<50% at Baseline).
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in the EuroQOL EQ-5D (Five Dimensions) Thermometer Score at Week 13 and Months 7, 10, 13, 16, and 25
Description: The EuroQol (EQ-5D) questionnaire is a 2-page, generic, preference-based quality of life measure comprised of a 5-item health status measure and a visual analogue scale (VAS) and is used to generate two scores: the utility score and the thermometer score The thermometer score is based on a vertical VAS. The VAS is designed like a thermometer scale on which the best health state the participant can imagine is referenced at 100, and the worst health state the participant can imagine is marked by 0. Based on how good or bad the current health state is, the participant is asked to draw a line across the thermometer scale. For example, a line drawn across 46 on the scale of 0 to 100 would be coded 46. A negative adjusted mean change from Baseline represents a worsening of quality of life. Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: Intent-to-Treat (ITT) Population: all randomized participants.
  Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 371 | 288
scores on a scale
  Week 13 | 1.35 (0.876) | 1.20 (0.993)
  Month 7: number analyzed (Participants) | 301 | 220
  Month 7 | 3.00 (0.929) | 1.69 (1.076)
  Month 10: number analyzed (Participants) | 225 | 179
  Month 10 | 3.68 (1.048) | 0.98 (1.179)
  Month 13: number analyzed (Participants) | 179 | 136
  Month 13 | 2.92 (1.194) | 2.49 (1.369)
  Month 16: number analyzed (Participants) | 127 | 87
  Month 16 | 3.30 (1.219) | 3.51 (1.451)
  Month 25: number analyzed (Participants) | 86 | 53
  Month 25 | 6.87 (1.534) | 1.71 (1.937)

15. Secondary Outcome: Change From Baseline in the EQ-5D (Five Dimensions) Utility Score at Week 13 and Months 7, 10, 13, 16, and 25
Description: The EQ-5D utility score captures health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety and/or depression. Participants indicated the level of perceived problems in each of the five dimensions on three levels: 1, no problems; 2, some problems; 3, an extreme problem. Unique health states were defined by combining response levels from each of the five dimensions. For example, state 11111 indicates no problem on any of the five dimensions, whereas state 11223 indicates no problems with mobility or self-care; some problems with performing usual activities, moderate pain/discomfort; and extreme anxiety/depression. Responses are typically converted into health utilities or valuations on a scale ranging from 0 (worst health) to 1 (perfect health). A negative adjusted mean change from Baseline represents a worsening of quality of life. Mean changes from Baseline were calculated via mixed model-repeated measures ANCOVA.
Time Frame: Baseline; Week 13; Months 7, 10, 13, 16, and 25
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 376 | 293
scores on a scale
  Week 13 | 0.00 (0.009) | -0.04 (0.010)
  Month 7: number analyzed (Participants) | 303 | 226
  Month 7 | 0.00 (0.010) | -0.04 (0.012)
  Month 10: number analyzed (Participants) | 228 | 181
  Month 10 | 0.01 (0.011) | -0.04 (0.012)
  Month 13: number analyzed (Participants) | 185 | 138
  Month 13 | 0.01 (0.011) | -0.01 (0.013)
  Month 16: number analyzed (Participants) | 129 | 87
  Month 16 | -0.00 (0.014) | 0.03 (0.017)
  Month 25: number analyzed (Participants) | 88 | 56
  Month 25 | 0.00 (0.016) | -0.02 (0.020)

16. Secondary Outcome: Number of Participants With the Indicated Grade 2, 3, and 4 On-therapy Adverse Events Occurring in >=10% of Participants in Either Treatment Arm
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were graded according to the Common Terminiology Criteria for Adverse Events (CTCAE), Version 4.0. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life threatening; Grade 5, death.
Time Frame: From the date of the first dose of study drug to the date of the last dose plus 28 days (average of 9.8 months for pazopanib and 12.6 months for placebo)
Population: All Treated Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 461 | 477
participants
  Hypertension, G2 | 52 | 95
  Hypertension, G3 | 25 | 139
  Hypertension, G4 | 0 | 0
  Diarrhoea, G2 | 22 | 97
  Diarrhoea, G3 | 5 | 38
  Diarrhoea, G4 | 0 | 1
  Nausea, G2 | 15 | 42
  Nausea, G3 | 0 | 4
  Nausea, G4 | 0 | 0
  Headache, G2 | 6 | 36
  Headache, G3 | 3 | 8
  Headache, G4 | 0 | 0
  Fatigue, G2 | 19 | 42
  Fatigue, G3 | 1 | 7
  Fatigue, G4 | 0 | 0
  Neutropenia, G2 | 17 | 51
  Neutropenia, G3 | 2 | 29
  Neutropenia, G4 | 2 | 3
  Dysgeusia, G2 | 0 | 16
  Dysgeusia, G3 | 0 | 0
  Dysgeusia, G4 | 0 | 0
  Abdominal pain, G2 | 21 | 26
  Abdominal pain, G3 | 5 | 5
  Abdominal pain, G4 | 0 | 0
  Alanine aminotransferase increased, G2 | 4 | 22
  Alanine aminotransferase increased, G3 | 0 | 24
  Alanine aminotransferase increased, G4 | 1 | 4
  Hair color changes, G2 | 0 | 13
  Hair color changes, G3 | 0 | 0
  Hair color changes, G4 | 0 | 0
  Decreased appetite, G2 | 2 | 19
  Decreased appetite, G3 | 0 | 1
  Decreased appetite, G4 | 0 | 0
  Vomiting, G2 | 8 | 21
  Vomiting, G3 | 1 | 4
  Vomiting, G4 | 0 | 0
  Aspartate aminotransferase increased, G2 | 3 | 22
  Aspartate aminotransferase increased, G3 | 0 | 10
  Aspartate aminotransferase increased, G4 | 1 | 3
  Arthralgia, G2 | 13 | 19
  Arthralgia, G3 | 3 | 5
  Arthralgia, G4 | 0 | 0
  Abdominal pain upper, G2 | 3 | 20
  Abdominal pain upper, G3 | 1 | 1
  Abdominal pain upper, G4 | 0 | 1
  Asthenia, G2 | 8 | 28
  Asthenia, G3 | 0 | 6
  Asthenia, G4 | 0 | 0
  Palmar-plantar erythrodysaesthesia syndrome, G2 | 2 | 42
  Palmar-plantar erythrodysaesthesia syndrome, G3 | 1 | 9
  Palmar-plantar erythrodysaesthesia syndrome, G4 | 0 | 0
  Thrombocytopenia, G2 | 1 | 15
  Thrombocytopenia, G3 | 1 | 6
  Thrombocytopenia, G4 | 2 | 3
  Hypothyroidism, G2 | 9 | 19
  Hypothyroidism, G3 | 0 | 0
  Hypothyroidism, G4 | 0 | 0
  Constipation, G2 | 20 | 12
  Constipation, G3 | 1 | 1
  Constipation, G4 | 0 | 0

17. Secondary Outcome: Number of Participants With the Indicated On-therapy Hematology Grade Shifts From Baseline Grade
Description: Hematology toxicities were graded according to the Common Terminiology Criteria for Adverse Events (CTCAE), Version 4.0. Grade refers to the severity of the toxicity. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life threatening; Grade 5, death. Participants with a missing Baseline grade were assumed to have a Baseline grade of 0. WBC=White blood cell.
Time Frame: as for outcome 16
Population: All Treated Population. Only those participants contributing toxicity data were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 456 | 466
participants
  Hemoglobin, Any grade increase | 44 | 68
  Hemoglobin, Increase to Grade 3 | 0 | 0
  Hemoglobin, Increase to Grade 4 | 0 | 0
  Lymphocytes, Any grade increase: number analyzed (Participants) | 453 | 461
  Lymphocytes, Any grade increase | 75 | 91
  Lymphocytes, Increase to Grade 3: number analyzed (Participants) | 453 | 461
  Lymphocytes, Increase to Grade 3 | 1 | 13
  Lymphocytes, Increase to Grade 4: number analyzed (Participants) | 453 | 461
  Lymphocytes, Increase to Grade 4 | 0 | 0
  Neutrophils, Any grade increase: number analyzed (Participants) | 455 | 462
  Neutrophils, Any grade increase | 80 | 236
  Neutrophils, Increase to Grade 3: number analyzed (Participants) | 455 | 462
  Neutrophils, Increase to Grade 3 | 2 | 44
  Neutrophils, Increase to Grade 4: number analyzed (Participants) | 455 | 462
  Neutrophils, Increase to Grade 4 | 0 | 5
  Platelets, Any grade increase: number analyzed (Participants) | 456 | 465
  Platelets, Any grade increase | 25 | 167
  Platelets, Increase to Grade 3: number analyzed (Participants) | 456 | 465
  Platelets, Increase to Grade 3 | 1 | 8
  Platelets, Increase to Grade 4: number analyzed (Participants) | 456 | 465
  Platelets, Increase to Grade 4 | 1 | 4
  WBC count, Any grade increase: number analyzed (Participants) | 456 | 465
  WBC count, Any grade increase | 77 | 236
  WBC count, Increase to Grade 3: number analyzed (Participants) | 456 | 465
  WBC count, Increase to Grade 3 | 0 | 11
  WBC count, Increase to Grade 4: number analyzed (Participants) | 456 | 465
  WBC count, Increase to Grade 4 | 0 | 1

18. Secondary Outcome: Number of Participants With the Indicated On-therapy Chemistry Grade Shifts From Baseline Grade
Description: Hematology toxicities were graded according to the Common Terminiology Criteria for Adverse Events (CTCAE), Version 4.0. Grade refers to the severity of the toxicity. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life threatening; Grade 5, death. Participants with a missing Baseline grade were assumed to have a Baseline grade of 0.
Time Frame: as for outcome 16
Population: All Treated Population. Only those participants contributing toxicity data were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 456 | 465
participants
  Albumin, Any grade increase: number analyzed (Participants) | 450 | 455
  Albumin, Any grade increase | 33 | 50
  Albumin, Increase to Grade 3: number analyzed (Participants) | 450 | 455
  Albumin, Increase to Grade 3 | 0 | 0
  Albumin, Increase to Grade 4: number analyzed (Participants) | 450 | 455
  Albumin, Increase to Grade 4 | 0 | 0
  Creatinine, Any grade increase | 27 | 42
  Creatinine, Increase to Grade 3 | 0 | 1
  Creatinine, Increase to Grade 4 | 0 | 0
  Hypercalcemia, Any grade increase: number analyzed (Participants) | 456 | 462
  Hypercalcemia, Any grade increase | 33 | 16
  Hypercalcemia, Increase to Grade 3: number analyzed (Participants) | 456 | 462
  Hypercalcemia, Increase to Grade 3 | 0 | 0
  Hypercalcemia, Increase to Grade 4: number analyzed (Participants) | 456 | 462
  Hypercalcemia, Increase to Grade 4 | 0 | 0
  Hyperglycemia, Any grade increase: number analyzed (Participants) | 446 | 453
  Hyperglycemia, Any grade increase | 117 | 128
  Hyperglycemia, Increase to Grade 3: number analyzed (Participants) | 446 | 453
  Hyperglycemia, Increase to Grade 3 | 10 | 2
  Hyperglycemia, Increase to Grade 4: number analyzed (Participants) | 446 | 453
  Hyperglycemia, Increase to Grade 4 | 0 | 0
  Hyperkalemia, Any grade increase: number analyzed (Participants) | 455 | 464
  Hyperkalemia, Any grade increase | 39 | 38
  Hyperkalemia, Increase to Grade 3: number analyzed (Participants) | 455 | 464
  Hyperkalemia, Increase to Grade 3 | 2 | 1
  Hyperkalemia, Increase to Grade 4: number analyzed (Participants) | 455 | 464
  Hyperkalemia, Increase to Grade 4 | 0 | 2
  Hypermagnesemia, Any grade increase: number analyzed (Participants) | 439 | 447
  Hypermagnesemia, Any grade increase | 11 | 20
  Hypermagnesemia, Increase to Grade 3: number analyzed (Participants) | 439 | 447
  Hypermagnesemia, Increase to Grade 3 | 1 | 6
  Hypermagnesemia, Increase to Grade 4: number analyzed (Participants) | 439 | 447
  Hypermagnesemia, Increase to Grade 4 | 1 | 0
  Hypernatremia, Any grade increase: number analyzed (Participants) | 455 | 463
  Hypernatremia, Any grade increase | 26 | 25
  Hypernatremia, Increase to Grade 3: number analyzed (Participants) | 455 | 463
  Hypernatremia, Increase to Grade 3 | 0 | 0
  Hypernatremia, Increase to Grade 4: number analyzed (Participants) | 455 | 463
  Hypernatremia, Increase to Grade 4 | 0 | 0
  Hypocalcemia, Any grade increase: number analyzed (Participants) | 456 | 462
  Hypocalcemia, Any grade increase | 21 | 52
  Hypocalcemia, Increase to Grade 3: number analyzed (Participants) | 456 | 462
  Hypocalcemia, Increase to Grade 3 | 0 | 2
  Hypocalcemia, Increase to Grade 4: number analyzed (Participants) | 456 | 462
  Hypocalcemia, Increase to Grade 4 | 0 | 0
  Hypoglycemia, Any grade increase: number analyzed (Participants) | 446 | 453
  Hypoglycemia, Any grade increase | 25 | 41
  Hypoglycemia, Increase to Grade 3: number analyzed (Participants) | 446 | 453
  Hypoglycemia, Increase to Grade 3 | 2 | 0
  Hypoglycemia, Increase to Grade 4: number analyzed (Participants) | 446 | 453
  Hypoglycemia, Increase to Grade 4 | 2 | 2
  Hypokalemia, Any grade increase: number analyzed (Participants) | 455 | 464
  Hypokalemia, Any grade increase | 31 | 40
  Hypokalemia, Increase to Grade 3: number analyzed (Participants) | 455 | 464
  Hypokalemia, Increase to Grade 3 | 1 | 2
  Hypokalemia, Increase to Grade 4: number analyzed (Participants) | 455 | 464
  Hypokalemia, Increase to Grade 4 | 1 | 0
  Hypomagnesemia, Any grade increase: number analyzed (Participants) | 439 | 447
  Hypomagnesemia, Any grade increase | 55 | 65
  Hypomagnesemia, Increase to Grade 3: number analyzed (Participants) | 439 | 447
  Hypomagnesemia, Increase to Grade 3 | 3 | 1
  Hypomagnesemia, Increase to Grade 4: number analyzed (Participants) | 439 | 447
  Hypomagnesemia, Increase to Grade 4 | 0 | 2
  Hyponatremia, Any grade increase: number analyzed (Participants) | 455 | 463
  Hyponatremia, Any grade increase | 37 | 45
  Hyponatremia, Increase to Grade 3: number analyzed (Participants) | 455 | 463
  Hyponatremia, Increase to Grade 3 | 5 | 9
  Hyponatremia, Increase to Grade 4: number analyzed (Participants) | 455 | 463
  Hyponatremia, Increase to Grade 4 | 0 | 0
  Phosphate, Any grade increase: number analyzed (Participants) | 409 | 401
  Phosphate, Any grade increase | 33 | 24
  Phosphate, Increase to Grade 3: number analyzed (Participants) | 409 | 401
  Phosphate, Increase to Grade 3 | 4 | 0
  Phosphate, Increase to Grade 4: number analyzed (Participants) | 409 | 401
  Phosphate, Increase to Grade 4 | 0 | 1

19. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Thyroid-stimulating Hormone (TSH) Elevations Above 5 Million Units Per Liter (MU/L)
Description: Participants were assessed for thyroid function abnormalities. Clinical hypothyroidism is defined as 5 <TSH <=10 MU/L and T4 <lower limit of normal (LLN).
Time Frame: as for outcome 16
Population: All Treated Population. Only those participants with any TSH above 5 MU/L were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 42 | 157
participants
  5 <TSH <=10 MU/L | 34 | 94
  10 <TSH <=20 MU/L | 4 | 36
  TSH >20 MU/L | 4 | 27

20. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study treatment up to 28 days after study drug discontinuation, for a maximum duration of 27 months. Deaths post treatment survival follow up were collected after the on treatment period, up to 96 months (8 years).
Time Frame: on-treatment: up to 27 months; post-treatment: up to 96 months (8 years).
Population: Treated set.
  One randomized patient in each treatment arm was excluded from the All Treated population because they did not receive treatment. The pazopanib group included 6 patients who were randomized to placebo but took at least one dose of pazopanib.
  Four patients (one in placebo, three in pazopanib) had missing death dates and therefore were treated as censored at the last contact date.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 mg
Number analyzed (Participants) | 461 | 477
participants
  All Treated Population | 461 | 477
  Total deaths | 252 | 245
  On-treatment Deaths - occurring less than or equal to 28 days from last dose | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 28 days post treatment, up to a maximum duration of approximately 25 months.
Groups:
- Pazopanib: Pazopanib
Arm/Group | Placebo | Pazopanib
All-Cause Mortality (participants affected / at risk) | 0/461 | 3/477
Serious Adverse Events (participants affected / at risk) | 51/461 | 121/477
Other Adverse Events (participants affected / at risk) | 381/461 | 462/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=461) | Pazopanib (N=477)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 2
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Fibrosis (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 4
Hernia (General disorders) | 1 | 2
Ill-defined disorder (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 9
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 3
Cytokine release syndrome (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Sarcoidosis (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 18
Aspartate aminotransferase increased (Investigations) | 0 | 7
Blood bilirubin increased (Investigations) | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 5
Liver function test abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant lymphoma unclassifiable low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ulcerated haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Transverse sinus thrombosis (Nervous system disorders) | 0 | 1
Device breakage (Product Issues) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 8
Hypertensive crisis (Vascular disorders) | 0 | 4
Lymphocele (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=461) | Pazopanib (N=477)
Leukopenia (Blood and lymphatic system disorders) | 5 | 44
Neutropenia (Blood and lymphatic system disorders) | 23 | 103
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 48
Hypothyroidism (Endocrine disorders) | 15 | 49
Abdominal pain (Gastrointestinal disorders) | 94 | 88
Abdominal pain upper (Gastrointestinal disorders) | 30 | 67
Constipation (Gastrointestinal disorders) | 72 | 38
Diarrhoea (Gastrointestinal disorders) | 79 | 252
Dyspepsia (Gastrointestinal disorders) | 17 | 24
Nausea (Gastrointestinal disorders) | 81 | 174
Stomatitis (Gastrointestinal disorders) | 7 | 27
Vomiting (Gastrointestinal disorders) | 39 | 71
Asthenia (General disorders) | 55 | 66
Fatigue (General disorders) | 66 | 133
Mucosal inflammation (General disorders) | 10 | 32
Urinary tract infection (Infections and infestations) | 33 | 32
Viral upper respiratory tract infection (Infections and infestations) | 24 | 27
Alanine aminotransferase increased (Investigations) | 25 | 73
Aspartate aminotransferase increased (Investigations) | 24 | 66
Blood alkaline phosphatase increased (Investigations) | 3 | 24
Blood bilirubin increased (Investigations) | 1 | 29
Blood thyroid stimulating hormone increased (Investigations) | 1 | 32
Neutrophil count decreased (Investigations) | 11 | 36
Platelet count decreased (Investigations) | 1 | 30
Decreased appetite (Metabolism and nutrition disorders) | 15 | 79
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 | 71
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 30
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 35
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 45
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 38
Dizziness (Nervous system disorders) | 22 | 26
Dysgeusia (Nervous system disorders) | 13 | 95
Headache (Nervous system disorders) | 70 | 135
Insomnia (Psychiatric disorders) | 27 | 24
Proteinuria (Renal and urinary disorders) | 8 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 31
Hair colour changes (Skin and subcutaneous tissue disorders) | 8 | 95
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 61
Rash (Skin and subcutaneous tissue disorders) | 22 | 42
Hot flush (Vascular disorders) | 29 | 23
Hypertension (Vascular disorders) | 87 | 256

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT00866697/SAP_000.pdf